CLINICAL TRIAL: NCT01573923
Title: Clinical Trial of Umbilical Mesenchymal Stem Cells Transplantation for Liver Cirrhosis-Phase I/II
Brief Title: Safety and Efficacy Study of Umbilical Mesenchymal Stem Cells for Liver Cirrhosis
Acronym: LC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alliancells Bioscience Corporation Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alliancells-2012-1
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2012-04

CONDITIONS: Liver Cirrhosis
Keywords: Umbilical Mesenchymal Stem Cells; Liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional therapy (Sham Comparator): only apply for conventional medical therapy without any cell therapy
  Interventions: Biological: Conventional therapy
- mesenchymal stem cells (Active Comparator): combination of conventional therapy with umbilical mesenchymal stem cells intravenous injection, (4x107/40ml, once per three months, four times in one year)
  Interventions: Biological: mesenchymal stem cells

INTERVENTIONS:
Biological: mesenchymal stem cells — Conventional therapy plus UC-MSC intravenous administration (4x107/40ml, once per three months, four times in one year)
  Arms: mesenchymal stem cells
Biological: Conventional therapy — Conventional therapy without cell therapy
  Arms: Conventional therapy

SUMMARY:
Liver cirrhosis and subsequent liver failure are leading causes of morbidity and mortality worldwide. Alcohol abuse and viral hepatitis are the most common causes of cirrhosis. Novel therapies are necessary to prevent or block the process of the disease. In this current prospective cohort, the investigators plan to organize four hospitals to determine the safety and efficacy of intravenous administration of umbilical mesenchymal stem cells in the treatment of patients with liver cirrhosis in next three years.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* aged 30-60 years
* clinical diagnosis of compensated or decompensated liver
* child-Pugh B/C (7-12 points)
* expecting lifetime is over three years

Exclusion Criteria:

* pregnant woman
* patient with severe vascular diseases
* patient with any organ failure
* patient with any tumors
* patient with HIV
* patient who has been transplanted
* patient treated with immunosuppressors
* patient for whom the follow-up is considered impossible
* patients with any disease or condition which the investigator or treating physician feels would interfere with the trial or the safety of the subject

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
survival time | 3-year follow up

SECONDARY OUTCOMES:
Serum markers regarding liver and kidney function | 0, 3, 6, 9 and 12 months
  liver functions：Albumin (ALB), Alanine aminotransferase (ALT), Aspartate Aminotransferase (AST), Prealbumin(PA), total bilirubin (TB), and direct bilirubin (DB) kidney function：Blood urea nitrogen (BUN), Urea (UA), and Crea (Cr)
Serum markers regarding lipid and sugar profile | 0, 3, 6, 9 and 12 months
  Total cholesterol (TC), high density lipoprotein cholesterol (HDL-C), low density lipoprotein cholesterol (LDL-C), triglycerides (TG), very low density lipoprotein cholesterol (VLDL-C), and Non-HDL-C; blood sugar;
Serum markers regarding cytokine profile | 0, 3, 6, 9 and 12 months
  IL-1β, IL-4, IL-6, IL-8, IL-10, IL-12(p40), IL-15, IL-17A, TNFα, TNFβ, IFN-γ, RANTES, TGFβ, lymphotactin, and C-reactive protein level (CRP)
Serum levels of Hepatitis B and C | 0, 3, 6, 9 and 12 months
  Serum levels of Hepatitis B and C
tolerance and the adverse events | 3-year follow up
  The classification for uncomfortable reaction is: 0, no discomfort; 1, slightly unwell, does not affect daily life; 2, moderate discomfort, affects daily life and work; 3, moderately unwell, significantly affects life, and bed rest; 4, severely unwell, life-threatening.
  A serious adverse event is defined as fatal, life threatening, permanently disabling, and tumors, particularly hepatocellular carcinoma.
Changes of any clinical symptoms | 3-year follow up
  abdominal distension, appetite, debilitation, and edema of lower limbs.

CONTACTS AND LOCATIONS:
Overall Officials: Xuetao Pei, MD,PhD, Study Chair — Chinese Industry and Innovative Technology Strategic Alliance of Stem Cells and Regenerative Medicine; Yongjun Liu, MD,PhD, Study Director — Alliancells Bioscience Corporation Limited; Mingyuan Wu, MD,PhD, Study Director — Eastern Union Stem Cell & Gene Engineering Co.,Ltd， Alliancells Bioscience Corporation Limited; Hanwei Li, MD,PhD, Principal Investigator — The 302 Hospital of Chinese People's Liberation Army; Liming Wang, MD, Principal Investigator — The 323 Hospital of Chinese People's Liberation Army; Xun Li, MD,PhD, Principal Investigator — LanZhou University; Liming Chen, MD,PhD, Principal Investigator — ongji Hospital of Tongji University; Jianwei Lu, MD, Principal Investigator — Tongji Hospital; Hui Shi, MD, Principal Investigator — The First People's Hospital of Lianyungang
Locations (6):
- China (6):
  - The 302 Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - the First Affiliated Hospital of Lanzhou University, Lanzhou, Gansu
  - Hainan BOAO Life infinity international anti-aging medical center, Qionghai, Hainan
  - The first people's hospital of Lianyungang, Lianyungang, Jiangsu
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - The 323 Hospital of Chinese People's Liberation Army, Xi’an, Shanxi